CLINICAL TRIAL: NCT00065741
Title: Botanical/Drug Interactions in HIV: Glucuronidation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21AT001376-01A1 (NIH)
Record Dates: First submitted 2003-07-31; First posted 2003-08-01 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2007-03

CONDITIONS: HIV Seronegativity
Keywords: Milk thistle; silymarin; piperine; glucarate; zidovudine; abacavir; mycophenolate mofetil; HIV; pharmacokinetics; interaction; glucuronidation; Healthy; Complementary Therapies
MeSH Terms: interventions — Silymarin

INTERVENTIONS:
Drug: silymarin

SUMMARY:
A series of clinical studies will be conducted in normal, healthy adult volunteers to evaluate the potential for alterations in the pharmacokinetics of anti HIV drugs when botanicals/nutriceuticals are given concurrently via the oral route. Both the drugs and botanicals are known to rely upon or to modulate, respectively, metabolism via glucuronidation.

DETAILED DESCRIPTION:
As per Brief Summary

ELIGIBILITY:
Inclusion criteria:

* Absence of HIV-1 infections

  * Body mass index less than or equal to 30 kg/m2 and weigh at least 50 kg.
* Laboratory values obtained within 7 days of study entry within normal range for healthy volunteers.
* Able to be compliant with dosing schedules and diary record keeping.
* Able to follow dietary restrictions associated with the protocol.
* Ability and willingness to provide informed consent
* All women of reproductive potential must have a negative pregnancy test
* All women of reproductive potential to use contraception methods as defined by protocol
* All study subjects (male and female) must agree to not participate in a conception process

Exclusion Criteria:

* History of any acute or chronic illness that requires current medical therapy including active gastrointestinal conditions that might interfere with drug absorption.
* History of hepatic, renal, cardiovascular, gastrointestinal diseases.
* Current gastrointestinal disturbance.
* Receipt of any prescribed or over the counter medication or ingested CAM during the 30 days prior to study entry except: Over the counter acetaminophen or ibuprofen at doses not exceeding package labeling guidelines.
* Any medical condition that, in the opinion of the investigator, would interfere with the subject's ability to participate in this protocol.
* Pregnancy or breastfeeding.
* Allergy/sensitivity to study agent(s) or their formulations.
* Active drug or alcohol abuse or dependence, which in the opinion of the investigator would interfere with adherence to study requirements or would endanger the subject's health while on study.
* Before entering the study, subjects must agree not to consume alcohol for 48 hours prior to PK sampling days.
* Participation in any investigational drug studies within 30 days prior to study entry and during study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2003-09; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Smith, PhD, Principal Investigator — School of Pharmacy, UNC Chapel Hill; David A Wohl, MD, Study Director — Department of Medicine, AIDS Clinical Trials Unit, University of North Carolina at Chapel Hill
Locations (1):
- General Clinical Research Center, Univiversity Of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States